CLINICAL TRIAL: NCT07317947
Title: The Effect of Lateral Crural Steal With Columellar Strut Graft on Nasal Tip Projection and Rotation in Primary Open Rhinoplasty
Brief Title: Lateral Crural Steal With Columellar Strut Graft in Primary Open Rhinoplasty
Acronym: LCS/CS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Elsaeed Habib, Plastic Surgery Resident, Kafrelsheikh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-725
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Rhinoplasty; Nasal Surgery; Aesthetic Outcomes
Keywords: Rhinoplasty; Lateral crural steal; Columellar strut; Rhinobase; Rhinoplasty Outcome Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Open Rhinoplasty (Experimental): Lateral crural steal with columellar strut graft will be done in patients undergoing Primary Open Rhinoplasty
  Interventions: Procedure: Lateral crural steal with columellar strut graft in Primary Open Rhinoplasty

INTERVENTIONS:
Procedure: Lateral crural steal with columellar strut graft in Primary Open Rhinoplasty — Patients undergo primary open rhinoplasty under general anesthesia. After local infiltration, an open approach is performed using an inverted-V transcolumellar incision with bilateral marginal incisions. The skin-soft tissue envelope is elevated in the supra-perichondrial plane. Dorsal deformities are corrected and septoplasty is performed with cartilage harvest. Vestibular skin is undermined and cephalic trimming of the lateral crura is carried out. Lateral crural steal is performed by advancing the medial end of the lateral crus 3-5 mm medially using transdomal sutures after defining the new dome position. A fixed columellar strut graft is inserted between the medial crura and secured to provide central tip support. Interdomal sutures are placed. No additional projection-enhancing grafts are used. Incisions are closed and internal and external nasal splints are applied.

SUMMARY:
The goal of this clinical trial is to assess the effect of Lateral crural steal with Columellar strut graft done in Primary Open Rhinoplasty and its long-term sustainability on nasal tip projection and nasal tip rotation.

DETAILED DESCRIPTION:
Rhinoplasty is one of the most commonly performed aesthetic procedures worldwide, with the nasal tip being the most challenging aspect of it. The nasal tip represents the most anterior projecting point of the nose and is formed by the junction of the medial and lateral crura of lower lateral cartilages.

Projection, rotation, and definition are key aspects to be controlled and achieved in the nasal tip surgery. Preservation of natural tip support is a fundamental requirement of a successful rhinoplasty.

Although excisional techniques can produce reductions in lobular width, long-term contour alterations are unpredictable and subject to stigmatic tip deformity. As a consequence, aggressive excision-based techniques are increasingly recognized as haphazard, unpredictable, and disproportionately prone to undesirable postoperative contour deformities.

The lateral crural steal (LCS) is a tissue-conservative technique of nasal tip refinement through relocation of domal apices. Hence, modifying nasal tip projection and rotation. However, the long-term stability of tip position with LCS alone can be variable. To enhance support and long-term maintenance of tip projection, a columellar strut graft -placed between the medial crura- acts as a central scaffold, unifying the nasal tip and helping to control the final nasal tip position.

The lateral crural steal technique alone can achieve improvements in nasal tip projection and rotation, but with weak medial crura, it can twist or compress down the medial crura, which will result in loss of tip height. So, in the technique being studied, combining the LCS with a columellar strut graft can provide both dynamic and static support to the nasal tip.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking primary rhinoplasty for aesthetic and/or functional indications.
* Presence of inadequate nasal tip projection and/or rotation suitable for correction using lateral crural steal with columellar strut graft.
* Ability to provide written informed consent and comply with follow-up visits.

Exclusion Criteria:

* History of prior nasal surgery.
* History of severe nasal trauma, altering cartilage architecture.
* Significant functional nasal obstruction requiring complex external nasal valve reconstruction.
* Patients with excessively wide alar base requiring alar base reduction involving vestibular sill excision (to prevent confounding on projection/rotation).
* Patients with facial skeletal or developmental abnormalities e.g. maxillary hypoplasia, maxillary prognathism, dentofacial deformities.
* Patients with psychiatric illness or Body Dysmorphic Disorder.
* Significant medical comorbidities contraindicating elective surgery or general anesthesia.
* Inability to provide informed consent or comply with follow-up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Nasal tip projection. | Analysis will be done preoperatively, immediate postoperatively, and at 6-month and 1-year postoperatively.
  Assessing nasal projection using Goode's ratio, which is the ratio between distance from the alar crease (vertical plane of the alar base) to the tip of the nose and distance from the nasion to the tip of the nose. The ideal ratio is between 0.55 to 0.60.
  Nasal tip projection will be assessed using Rhinobase® software developed by Apaydin et al (2009), which is a software for rhinoplasty that enables standardized photographic analysis, facilitates precise anthropometric measurements, and provides objective documentation of pre- and postoperative nasal parameters.
Nasal tip rotation | Analysis will be done preoperatively, immediate postoperatively, and at 6-month and 1-year postoperatively.
  Assessing nasal tip rotation through measuring the Nasolabial angle which is the angle formed at the junction of the columella and a line drawn from the subnasale to the labrale superius, and the Nasofacial angle which is the angle between the nasal dorsum and the facial plane (glabella to pogonion).
  Nasal tip rotation will be assessed using Rhinobase® software developed by Apaydin et al (2009), which is a software for rhinoplasty that enables standardized photographic analysis, facilitates precise anthropometric measurements, and provides objective documentation of pre- and postoperative nasal parameters.

SECONDARY OUTCOMES:
Patient's satisfaction | The questionnaire will be conducted pre-operatively (as a baseline), 3-month and 1-year postoperatively.
  Assessing patient satisfaction through Rhinoplasty Outcome Evaluation (ROE) Questionnaire; which is a six-question questionnaire used to assess satisfaction with aesthetic and functional results after Rhinoplasty. Each of the six items is scored on a 0-4 scale, with 0 representing the most negative response and 4 representing the most positive response. Therefore, the total score can vary from 0 to 24. In order to facilitate the comprehension of the results, the total score can be divided by 24 and multiplied by 100, so that the score can vary from 0 to 100 %. So, 24 points or 100 % means the most patient satisfaction. It's originally piloted by Alsarraf (2000). The questionnaire has an Arabic-translated version done by Alharethy S, et al. (2021) that will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Safwat Adel Hegazy, Study Director — Kafrelsheikh University; Khaled Ahmed Ismail, Study Chair — Kafrelsheikh University
Locations (1):
- Kafrelsheikh University Hospital, Kafr ash Shaykh, Egypt

REFERENCES:
- [Background] Mulafikh DS, Alharethy SE, Alqabbani AA, Mesallam TA. Validation and clinical application of the Arabic rhinoplasty outcomes evaluation questionnaire. Saudi Med J. 2021 Jun;42(6):655-659. doi: 10.15537/smj.2021.42.6.20210038. PMID 34078728
- [Background] Alsarraf R. Outcomes research in facial plastic surgery: a review and new directions. Aesthetic Plast Surg. 2000 May-Jun;24(3):192-7. doi: 10.1007/s002660010031. PMID 10890946
- [Background] Apaydin F, Akyildiz S, Hecht DA, Toriumi DM. Rhinobase: a comprehensive database, facial analysis, and picture-archiving software for rhinoplasty. Arch Facial Plast Surg. 2009 May-Jun;11(3):209-11. doi: 10.1001/archfacial.2009.35. No abstract available. PMID 19451458
- [Background] Cetiner H. The Effect of Anchoring the Columellar Strut Graft to the Lateral Crural Steal Suture in Patients With a Low Nasal Tip: A New Technique. J Craniofac Surg. 2019 Mar/Apr;30(2):437-441. doi: 10.1097/SCS.0000000000005110. PMID 30614999
- [Background] Davis RE. Lateral crural tensioning for refinement of the wide and underprojected nasal tip: rethinking the lateral crural steal. Facial Plast Surg Clin North Am. 2015 Feb;23(1):23-53. doi: 10.1016/j.fsc.2014.09.003. PMID 25430927
- [Background] Kridel RW, Konior RJ, Shumrick KA, Wright WK. Advances in nasal tip surgery. The lateral crural steal. Arch Otolaryngol Head Neck Surg. 1989 Oct;115(10):1206-12. doi: 10.1001/archotol.1989.01860340060018. PMID 2789776
- [Background] Sepehr A, Alexander AJ, Chauhan N, Chan H, Adamson PA. Cephalic positioning of the lateral crura: implications for nasal tip-plasty. Arch Facial Plast Surg. 2010 Nov-Dec;12(6):379-84. doi: 10.1001/archfacial.2010.87. PMID 21079114
- [Background] Toriumi DM. New concepts in nasal tip contouring. Arch Facial Plast Surg. 2006 May-Jun;8(3):156-85. doi: 10.1001/archfaci.8.3.156. PMID 16702528
- [Background] Westreich RW, Lawson W. The tripod theory of nasal tip support revisited: the cantilevered spring model. Arch Facial Plast Surg. 2008 May-Jun;10(3):170-9. doi: 10.1001/archfaci.10.3.170. PMID 18490543
- [Background] Moubayed SP, Abou Chacra Z, Kridel RW, Ahmarani C, Rahal A. Precise anatomical study of rhinoplasty: description of a novel method and application to the lateral crural steal. JAMA Facial Plast Surg. 2014 Jan-Feb;16(1):25-30. doi: 10.1001/jamafacial.2013.1416. PMID 24177341